CLINICAL TRIAL: NCT03698123
Title: Performance Nutrition for Residents and Fellows Working Overnight Shifts: A Pilot Study
Brief Title: Performance Nutrition for Residents and Fellows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Medical Association (Other)
Responsible Party: Principal Investigator, Tait Shanafelt, Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 45690
Record Dates: First submitted 2018-09-25; First posted 2018-10-05 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Physician Well-being; Cognitive Function; Diet Modification; Diet Habit; Shift-Work Related Sleep Disturbance; Sleep Deprivation
Keywords: Nutrition; Physician well-being; Cognitive performance; Sleepiness; Shift-work
MeSH Terms: conditions — Feeding Behavior; Sleep Deprivation; Sleepiness | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Study participants will participate in the study 3 nights with one control night and two dietary interventions nights.The order of the 2 dietary intervention groups will be randomized per block.
  There are two possible combinations and the order will be randomized using a computer-generated random-number sequence. There will be at least a 24-hour wash-out period between study nights to minimize the carry-over effects of the cross-over design as well as learning effects of the computerized cognitive tests.
  A: Control- no intervention, B: intervention 1 arm, C: Intervention 2 The order of the blocks will be randomized. block a: A, B, C block b: A, C, B
Masking Description: Researchers analyze the data will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Modification (Experimental): On the first night of the study, participants can eat and drink as they normally would (no dietary intervention). On second and third nights participants will be provided meals, snacks and drinks with specific macronutrient composition, encouraged to only eat and drink study meals, snacks and drinks, and to avoid eating after 10:00 hours. The composition of the study foods and drinks on nights 2 and 3 will be different.
  Interventions: Other: Dietary Modification

INTERVENTIONS:
Other: Dietary Modification — Participants will be provided with meals, snacks and drinks with specific macronutrient compositions and encouraged to only eat and drink study meals, snacks and drinks and to avoid eating after 10:00 hours.

SUMMARY:
Currently, residents commonly experience dehydration and poor nutrition during nighttime duty hours as a result of heavy work load, lack of time to take nutrition and hydration breaks, or limited or no access to healthy food and drinks which may affect residents' work performance. The goal of this study is to compare the effects of two different meal compositions with no typical dietary practices (existing conditions) on work performance of the on-call residents during night shifts.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of dietary modifications on resident physicians' work performance during night shifts.

Specific objectives are:

1. To assess the effects of macronutrient composition of the test meals on cognitive performance, self-reported sleepiness and fatigue of resident physicians during night-time duty.
2. To compare to no intervention, the effects of providing meals before 22:00 hours, and only providing chewing gum, tea, coffee and water onwards to on-call residents, on cognitive performance, self-reported sleepiness and fatigue of resident physicians during night-time duty.

ELIGIBILITY:
Inclusion Criteria:

* All residents and fellows performing in hospital overnight work
* Must be able to eat plant source foods (e.g. soy, nuts, seeds) and animal source foods (e.g. meat, eggs, dairy products)

Exclusion Criteria:

* Food allergies or sensitivities
* Prior anaphylactic reaction to food
* Strict dietary restrictions (e.g. vegan, gluten free)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-05-11 (Actual); Study Completion 2019-05-11 (Actual)

PRIMARY OUTCOMES:
Difference in Motor Praxis scores between conditions | Two time points (beginning and end of night shifts) on each night for a total of 3 nights
  Motor Praxis is a validated neurocognitive test that assesses sensory-motor speed. This test takes approximately 30 seconds to complete and will be measured at two time points (beginning and end of each night shift) in each of the 3 conditions . Differences in accuracy (percentage of correct responses, a higher percentage is better), duration (in milliseconds, lower duration is better), reaction time (in milliseconds, lower reaction time is better) and composite scores (0-1000, higher score is better) will be reported and compared.
Difference in Fractal 2-Back between conditions | Two time points (beginning and end of night shifts) on each night for a total of 3 nights
  Fractal 2-Back is a validated neurocognitive test that assess working memory. This test takes approximately 2 minutes to complete and will be measured at two time points (beginning and end of each night shift) in each of the 3 conditions. Differences in reaction time (in milliseconds, lower reaction time is better) , accuracy (percentage of correct responses, a higher percentage is better) and composite scores (0-1000, higher score is better) will be reported and compared.
Difference in Balloon Analog Risk between conditions | Two time points (beginning and end of night shifts) on each night for a total of 3 nights
  Balloon Analog Risk is a validated neurocognitive test that assess risk decision making. This test takes approximately 2 minutes to complete and will be measured at two time points (beginning and end of each night shift) in each of the 3 conditions. Differences in risk propensity (higher scores indicative of greater risk-taking propensity), duration (in milliseconds, lower reaction time is better) and composite scores (0-1000, higher score is better) will be reported and compared.
Difference in Psychomotor vigilance test between conditions | Two time points (beginning and end of night shifts) on each night for a total of 3 nights
  Psychomotor vigilance test is a validated neurocognitive test that assess vigilant attention. This test takes approximately 3 minutes to complete will be measured at two time points (beginning and end of each night shift) in each of the 3 conditions. Differences in reaction time (in milliseconds, lower reaction time is better), lapses (number, less is better) and composite scores measured (0-1000, higher score is better) will be reported and compared.

SECONDARY OUTCOMES:
Difference in Degree of sleepiness between conditions | Two time points (beginning and end of night shifts) on each night for a total of 3 nights
  Will use validated Stanford Sleepiness Scale (SSS) developed by William C. Dement, M.D., Ph.D. SSS a self-rating scale used to quantify progressive steps in sleepiness at a certain point in time. It is a seven-point Likert-type scale ranging from "feeling active, vital alert, or wide awake" (score = 1) to "no longer fighting sleep, sleep onset soon and having dream-like thoughts" (score = 7). Selected scores by the participants will be reported each time. This test takes approximately 15 seconds to complete. Differences in degree of sleepiness measured at two time points (beginning and end of each night shift) in each of the 3 conditions will be reported and compared.

OTHER OUTCOMES:
Difference in Work Exhaustion between conditions | Two time points (beginning and end of night shifts) on each night for a total of 3 nights
  Work Exhaustion scale, developed and modified by Mickey Trockel MD, PhD, to explore the degree of work related fatigue in residents and fellows. It has 4 questions with a 5 point Likert scale ranging from not at all to extremely. This test takes approximately 30 second to complete. The total score is the average scores of the 4 items and falls between 0 and 4. Scores equal to higher than 1.33 indicate work-related fatigue. Differences in Work Exhaustion scores measured at two time points (beginning and end of each night shift) in each of the 3 conditions will be reported and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Tait D Shanafelt, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
This data is strictly confidential and to protect the privacy of our study participants we will not be sharing the results.

REFERENCES:
- [Background] Rimmer A. Urgent action is needed to manage doctors' fatigue, says BMA. BMJ. 2018 Jan 9;360:k127. doi: 10.1136/bmj.k127. No abstract available. PMID 29317408
- [Background] Hamidi MS, Boggild MK, Cheung AM. Running on empty: a review of nutrition and physicians' well-being. Postgrad Med J. 2016 Aug;92(1090):478-81. doi: 10.1136/postgradmedj-2016-134131. Epub 2016 May 23. PMID 27215232
- [Background] Gupta CC, Dorrian J, Grant CL, Pajcin M, Coates AM, Kennaway DJ, Wittert GA, Heilbronn LK, Della Vedova CB, Banks S. It's not just what you eat but when: The impact of eating a meal during simulated shift work on driving performance. Chronobiol Int. 2017;34(1):66-77. doi: 10.1080/07420528.2016.1237520. Epub 2016 Oct 13. PMID 27736177
- [Background] Paech GM, Banks S, Pajcin M, Grant C, Johnson K, Kamimori GH, Vedova CB. Caffeine administration at night during extended wakefulness effectively mitigates performance impairment but not subjective assessments of fatigue and sleepiness. Pharmacol Biochem Behav. 2016 Jun;145:27-32. doi: 10.1016/j.pbb.2016.03.011. Epub 2016 Apr 7. PMID 27061779
- [Background] Grant CL, Dorrian J, Coates AM, Pajcin M, Kennaway DJ, Wittert GA, Heilbronn LK, Vedova CD, Gupta CC, Banks S. The impact of meal timing on performance, sleepiness, gastric upset, and hunger during simulated night shift. Ind Health. 2017 Oct 7;55(5):423-436. doi: 10.2486/indhealth.2017-0047. Epub 2017 Jul 25. PMID 28740034
- [Background] Reyner LA, Wells SJ, Mortlock V, Horne JA. 'Post-lunch' sleepiness during prolonged, monotonous driving - effects of meal size. Physiol Behav. 2012 Feb 28;105(4):1088-91. doi: 10.1016/j.physbeh.2011.11.025. Epub 2011 Dec 6. PMID 22155490
- [Background] Attuquayefio T, Stevenson RJ, Oaten MJ, Francis HM. A four-day Western-style dietary intervention causes reductions in hippocampal-dependent learning and memory and interoceptive sensitivity. PLoS One. 2017 Feb 23;12(2):e0172645. doi: 10.1371/journal.pone.0172645. eCollection 2017. PMID 28231304
- [Background] El-Sharkawy AM, Bragg D, Watson P, Neal K, Sahota O, Maughan RJ, Lobo DN. Hydration amongst nurses and doctors on-call (the HANDS on prospective cohort study). Clin Nutr. 2016 Aug;35(4):935-42. doi: 10.1016/j.clnu.2015.07.007. Epub 2015 Jul 16. PMID 26216194
- [Result] Makowski MS, Trockel MT, Menon NK, Wang H, Katznelson L, Shanafelt TD. Performance Nutrition for Physician Trainees Working Overnight Shifts: A Randomized Controlled Trial. Acad Med. 2022 Mar 1;97(3):426-435. doi: 10.1097/ACM.0000000000004509. PMID 34753859